CLINICAL TRIAL: NCT00833573
Title: National Survey on GERD Patients (Adults and Children)
Acronym: RGO à trav
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Alain Castaigne, Medical Director, AstraZeneca Pharmaceuticals
Other Study IDs: NIS-GFR-DUM-2008/2
Record Dates: First submitted 2009-01-30; First posted 2009-02-02 (Estimated); Last update posted 2009-11-17 (Estimated); Status verified 2009-11

CONDITIONS: GERD (Gastroesophageal Reflux Disease)
Keywords: GERD digestive expression; ages
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: For GP : the first 3 consecutive adult patients and the first children seen during the GP's visit with a diagnosis of GERD.
- 2: For Paediatrics : the first 2 consecutive children seen during the Paediatric's visit with a diagnosis of GERD.

SUMMARY:
To describe GERD digestive expression according to ages: - children (from 0 to 23 months) and (24 months and more)- adults (from 18 to 29 years old), (from 30 to 39 years old), (from 40 to 49 years old), (from 50 to 59 years old), (more than 60 years old)

ELIGIBILITY:
Inclusion Criteria:

* Adults : - Male or female > or = 18 years old - With at least one GERD typical clinical sign (pyrosis and / or acid regurgitations).- Not receiving any GERD treatment within the 3 previous months.
* Children :- Male or female < 18 years old - With GERD digestive clinical signs during the consultation (receiving treatment or not)- Whose parents or legal guardian gave oral approval to the child participation in the survey.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: For GP : the first 3 consecutive adult patients and the first children seen during the GP's visit with a diagnosis of GERD.For Paediatrics : the first 2 consecutive children seen during the Paediatric's visit with a diagnosis of GERD.
Sampling Method: Probability Sample
Enrollment: 4400 (Estimated)
Dates: Start 2009-01; Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
To describe GERD digestive expression according to ages: - children (from 0-23 months) and (24 months and more)- adults (from 18-29 years old), (from 30-39 years old), (from 40-49 years old), (from 50-59 years old), (more than 60 years old) | once

CONTACTS AND LOCATIONS:
Overall Officials: Alain Castaigne, Study Director — AstraZeneca
Locations (1053):
- France (1053):
  - Research Site, Abbaretz
  - Research Site, Abbeville
  - Research Site, Acheux-en-Amiénois
  - Research Site, Achicourt
  - Research Site, Adriers
  - Research Site, Agen
  - Research Site, Aigrefeuille-sur-Maine
  - Research Site, Aire-sur-l'Adour
  - Research Site, Aire-sur-la-Lys
  - Research Site, Airvault
  - Research Site, Aix-en-Othe
  - Research Site, Aix-en-Provence
  - Research Site, Aix-les-Bains
  - Research Site, Aizenay
  - Research Site, Ajaccio
  - Research Site, Albi
  - Research Site, Alençon
  - Research Site, Alès
  - Research Site, Alfortville
  - Research Site, Allonnes
  - Research Site, Althen-des-Paluds
  - Research Site, Ambès
  - Research Site, Ambillou-Château
  - Research Site, Amboise
  - Research Site, Amiens
  - Research Site, Andernos-les-Bains
  - Research Site, Angers
  - Research Site, Anglet
  - Research Site, Angoulême
  - Research Site, Annecy
  - Research Site, Annecy-le-Vieux
  - Research Site, Annezin
  - Research Site, Annonay
  - Research Site, Antibes
  - Research Site, Apremont
  - Research Site, Arc-et-Senans
  - Research Site, Arcachon
  - Research Site, Ardentes
  - Research Site, Argences
  - Research Site, Argentat
  - Research Site, Argenteuil
  - Research Site, Argenton-sur-Creuse
  - Research Site, Arnèke
  - Research Site, Arpajon
  - Research Site, Arques-la-Bataille
  - Research Site, Arras
  - Research Site, Ars
  - Research Site, Ars-sur-Moselle
  - Research Site, Art-sur-Meurthe
  - Research Site, Artenay
  - Research Site, Arudy
  - Research Site, Arzon
  - Research Site, Asnières-sur-Seine
  - Research Site, Aubenas
  - Research Site, Aubervilliers
  - Research Site, Auby
  - Research Site, Aucamville
  - Research Site, Auch
  - Research Site, Aulnay-sous-Bois
  - Research Site, Auray
  - Research Site, Aurec-sur-Loire
  - Research Site, Aussonne
  - Research Site, Auxerre
  - Research Site, Auxi-le-Château
  - Research Site, Auxon
  - Research Site, Auxonne
  - Research Site, Avelin
  - Research Site, Avesnelles
  - Research Site, Avignon
  - Research Site, Avord
  - Research Site, Avricourt
  - Research Site, Bagneux
  - Research Site, Bagnères-de-Luchon
  - Research Site, Bagnolet
  - Research Site, Bagnols-sur-Cèze
  - Research Site, Baignes Ste Radegonde
  - Research Site, Baillargues
  - Research Site, Bailleul
  - Research Site, Bais
  - Research Site, Balbigny
  - Research Site, Bandol
  - Research Site, Banyuls de la Marenda
  - Research Site, Barbentane
  - Research Site, Barbezieux-Saint-Hilaire
  - Research Site, Bardos
  - Research Site, Bassens
  - Research Site, Bastia
  - Research Site, Baugé
  - Research Site, Baulon
  - Research Site, Bayeux
  - Research Site, Bayonne
  - Research Site, Bâgé-le-Châtel
  - Research Site, Beaucouzé
  - Research Site, Beaumesnil
  - Research Site, Beaumont
  - Research Site, Beaumont-de-Pertuis
  - Research Site, Beaumont-Hague
  - Research Site, Beautor
  - Research Site, Beauvais
  - Research Site, Beauvoir-sur-Niort
  - Research Site, Belleville-sur-Meuse
  - Research Site, Bergerac
  - Research Site, Bernay
  - Research Site, Bersée
  - Research Site, Besançon
  - Research Site, Bécon-les-Granits
  - Research Site, Bégard
  - Research Site, Bérat
  - Research Site, Béruges
  - Research Site, Béthisy-Saint-Pierre
  - Research Site, Béthune
  - Research Site, Béville-le-Comte
  - Research Site, Béziers
  - Research Site, Biarritz
  - Research Site, Bignan
  - Research Site, Biscarrosse
  - Research Site, Bischheim
  - Research Site, Biver
  - Research Site, Bize-Minervois
  - Research Site, Blagnac
  - Research Site, Blangy-sur-Bresle
  - Research Site, Blanquefort
  - Research Site, Blaye
  - Research Site, Blénod-lès-Pont-à-Mousson
  - Research Site, Bobigny
  - Research Site, Bohain-en-Vermandois
  - Research Site, Boiscommun
  - Research Site, Bondues
  - Research Site, Bordeaux
  - Research Site, Bords
  - Research Site, Bormes-les-Mimosas
  - Research Site, Bosmie-l'Aiguille
  - Research Site, Bouc-Bel-Air
  - Research Site, Boucau
  - Research Site, Bouliac
  - Research Site, Boulogne-Billancourt
  - Research Site, Boulogne-sur-Gesse
  - Research Site, Boulogne-sur-Mer
  - Research Site, Bourbriac
  - Research Site, Bourg-en-Bresse
  - Research Site, Bourg-la-Reine
  - Research Site, Bourgoin
  - Research Site, Bourron-Marlotte
  - Research Site, Bracieux
  - Research Site, Braine
  - Research Site, Bram
  - Research Site, Brantôme
  - Research Site, Brax
  - Research Site, Bresles
  - Research Site, Brest
  - Research Site, Bretignolles-sur-Mer
  - Research Site, Briançon
  - Research Site, Brienne-le-Château
  - Research Site, Brienon-sur-Armançon
  - Research Site, Brignais
  - Research Site, Brioude
  - Research Site, Bruay-la-Buissière
  - Research Site, Brunstatt
  - Research Site, Bruyères
  - Research Site, Bruz
  - Research Site, Bry-sur-Marne
  - Research Site, Bubry
  - Research Site, Bures-sur-Yvette
  - Research Site, Burie
  - Research Site, Cachan
  - Research Site, Caen
  - Research Site, Cagnes-sur-Mer
  - Research Site, Cahuzac-sur-Vère
  - Research Site, Caluire-et-Cuire
  - Research Site, Cambrai
  - Research Site, Campagne-lès-Hesdin
  - Research Site, Candé
  - Research Site, Canet-en-Roussillon
  - Research Site, Cannes
  - Research Site, Cannes La Bocca
  - Research Site, Cany-Barville
  - Research Site, Capbreton
  - Research Site, Capdenac-Gare
  - Research Site, Carbon-Blanc
  - Research Site, Carcassonne
  - Research Site, Carentan
  - Research Site, Carhaix-Plouguer
  - Research Site, Carrières-sur-Seine
  - Research Site, Carros
  - Research Site, Carrouges
  - Research Site, Carry-le-Rouet
  - Research Site, Carvin
  - Research Site, Cassis
  - Research Site, Casteljaloux
  - Research Site, Castelnau-de-Guers
  - Research Site, Castelnaudary
  - Research Site, Castets-en-Dorthe
  - Research Site, Castres
  - Research Site, Catillon-sur-Sambre
  - Research Site, Catus
  - Research Site, Caulnes
  - Research Site, Cavaillon
  - Research Site, Cavignac
  - Research Site, Celles-sur-Plaine
  - Research Site, Cesson
  - Research Site, Cesson-Sévigné
  - Research Site, Cestas
  - Research Site, Cénac
  - Research Site, Chabris
  - Research Site, Chalais
  - Research Site, Chalonnes-sur-Loire
  - Research Site, Chamalières
  - Research Site, Chambéry
  - Research Site, Chambon-sur-Voueize
  - Research Site, Chamonix
  - Research Site, Champagne-sur-Seine
  - Research Site, Champagnole
  - Research Site, Champcueil
  - Research Site, Champeaux
  - Research Site, Champenoux
  - Research Site, Champigny-sur-Marne
  - Research Site, Champniers
  - Research Site, Champs-sur-Marne
  - Research Site, Chantepie
  - Research Site, Chantilly
  - Research Site, Chaource
  - Research Site, Charleville-Mézières
  - Research Site, Charmont-sous-Barbuise
  - Research Site, Chartres
  - Research Site, Chasseneuil-sur-Bonnieure
  - Research Site, Chauché
  - Research Site, Châlette-sur-Loing
  - Research Site, Châlons-en-Champagne
  - Research Site, Château-Arnoux-Saint-Auban
  - Research Site, Château-sur-Epte
  - Research Site, Châteaubriant
  - Research Site, Châteaugay
  - Research Site, Châteaumeillant
  - Research Site, Châteauneuf-en-Thymerais
  - Research Site, Châteauneuf-sur-Cher
  - Research Site, Châteauroux
  - Research Site, Châtel-Censoir
  - Research Site, Châtenay-Malabry
  - Research Site, Châtillon-sur-Marne
  - Research Site, Cherbourg Octeville Cedex
  - Research Site, Chinon
  - Research Site, Ciboure
  - Research Site, Cinq-Mars-la-Pile
  - Research Site, Claix
  - Research Site, Clamart
  - Research Site, Clermont-Ferrand
  - Research Site, Clichy
  - Research Site, Clichy-sous-Bois
  - Research Site, Clouange
  - Research Site, Cluny
  - Research Site, Coincy
  - Research Site, Colmar
  - Research Site, Colomars
  - Research Site, Colombes
  - Research Site, Combloux
  - Research Site, Combs-la-Ville
  - Research Site, Commentry
  - Research Site, Compiègne
  - Research Site, Concarneau
  - Research Site, Conty
  - Research Site, Coquelles
  - Research Site, Cornebarrieu
  - Research Site, Corseul
  - Research Site, Coudekerque-Branche
  - Research Site, Couffé
  - Research Site, Coulanges-lès-Nevers
  - Research Site, Coulommiers
  - Research Site, Courbevoie
  - Research Site, Cournon-d'Auvergne
  - Research Site, Courrières
  - Research Site, Courseulles-sur-Mer
  - Research Site, Coutouvre
  - Research Site, Couze-et-Saint-Front
  - Research Site, Coye-la-Forêt
  - Research Site, Creutzwald
  - Research Site, Creysse
  - Research Site, Crèvecœur-le-Grand
  - Research Site, Crécy-sur-Serre
  - Research Site, Créteil
  - Research Site, Criel-sur-Mer
  - Research Site, Criquetot-l'Esneval
  - Research Site, Croix
  - Research Site, Cros-de-Cagnes
  - Research Site, Crosne
  - Research Site, Cuers
  - Research Site, Cugnaux
  - Research Site, Cusset
  - Research Site, Dambach-la-Ville
  - Research Site, Daoulas
  - Research Site, Daux
  - Research Site, Decize
  - Research Site, Derval
  - Research Site, Décines-Charpieu
  - Research Site, Dieppe
  - Research Site, Dijon
  - Research Site, Dinard
  - Research Site, Divion
  - Research Site, Dole
  - Research Site, Domfront
  - Research Site, Domont
  - Research Site, Dompierre-sur-Besbre
  - Research Site, Donges
  - Research Site, Dossenheim-sur-Zinsel
  - Research Site, Douai
  - Research Site, Dozulé
  - Research Site, Drancy
  - Research Site, Droué
  - Research Site, Drumettaz
  - Research Site, Dugny-sur-Meuse
  - Research Site, Dunkirk
  - Research Site, Eckwersheim
  - Research Site, Elbeuf
  - Research Site, Embrun
  - Research Site, Enghien-les-Bains
  - Research Site, Entrammes
  - Research Site, Envermeu
  - Research Site, Erbalunga
  - Research Site, Ergué-Gabéric
  - Research Site, Escaudœuvres
  - Research Site, Eschau
  - Research Site, Estaires
  - Research Site, Estivareilles
  - Research Site, Estrablin
  - Research Site, Estrées-Saint-Denis
  - Research Site, Eyragues
  - Research Site, Eysines
  - Research Site, Écouflant
  - Research Site, Épieds-en-Beauce
  - Research Site, Épinal
  - Research Site, Épinay-sous-Sénart
  - Research Site, Épinay-sur-Orge
  - Research Site, Épinay-sur-Seine
  - Research Site, Équeurdreville-Hainneville
  - Research Site, Étaules
  - Research Site, Étretat
  - Research Site, Étupes
  - Research Site, Évreux
  - Research Site, Ézy-sur-Eure
  - Research Site, Fayence
  - Research Site, Fegersheim
  - Research Site, Fenouillet
  - Research Site, Fermanville
  - Research Site, Ferrières-en-Gâtinais
  - Research Site, Feurs
  - Research Site, Feyzin
  - Research Site, Figeac
  - Research Site, Firmi
  - Research Site, Firminy
  - Research Site, Fitz-James
  - Research Site, Flavin
  - Research Site, Fleury-les-Aubrais
  - Research Site, Fleury-sur-Orne
  - Research Site, Floirac
  - Research Site, Florac
  - Research Site, Folembray
  - Research Site, Fondettes
  - Research Site, Fontaine
  - Research Site, Fontaine-au-Pire
  - Research Site, Fontaine-lès-Dijon
  - Research Site, Fontenay-le-Comte
  - Research Site, Fontenay-le-Fleury
  - Research Site, Fontenay-sous-Bois
  - Research Site, Fontès
  - Research Site, Forges-les-Eaux
  - Research Site, Fougères
  - Research Site, Fouras
  - Research Site, Fourchambault
  - Research Site, Foussais-Payré
  - Research Site, Franconville
  - Research Site, Fréjus
  - Research Site, Froissy
  - Research Site, Fromentine
  - Research Site, Ganges
  - Research Site, Gap
  - Research Site, Garéoult
  - Research Site, Garges-lès-Gonesse
  - Research Site, Gelos
  - Research Site, Genillé
  - Research Site, Genlis
  - Research Site, Gentilly
  - Research Site, Ger
  - Research Site, Gif-sur-Yvette
  - Research Site, Gironde-sur-Dropt
  - Research Site, Givet
  - Research Site, Givors
  - Research Site, Gondrecourt-le-Château
  - Research Site, Gourdon
  - Research Site, Gournay-en-Bray
  - Research Site, Grand-Fougeray
  - Research Site, Granville
  - Research Site, Grenoble
  - Research Site, Grièges
  - Research Site, Grignols
  - Research Site, Guenrouet
  - Research Site, Guesnain
  - Research Site, Guignicourt
  - Research Site, Guipry
  - Research Site, Guissény
  - Research Site, Guîtres
  - Research Site, Gurgy
  - Research Site, Hagondange
  - Research Site, Haguenau
  - Research Site, Haillicourt
  - Research Site, Hanvec
  - Research Site, Harnes
  - Research Site, Hazebrouck
  - Research Site, Hendaye
  - Research Site, Hennebont
  - Research Site, Hesdin
  - Research Site, Hillion
  - Research Site, Hombourg-Haut
  - Research Site, Hondeghem
  - Research Site, Hundling
  - Research Site, Huriel
  - Research Site, Hyères
  - Research Site, Illiers-Combray
  - Research Site, Inchy
  - Research Site, Ingré
  - Research Site, Is-sur-Tille
  - Research Site, Isle
  - Research Site, Issoire
  - Research Site, Issoudun
  - Research Site, Issy-les-Moulineaux
  - Research Site, Istres
  - Research Site, Ivry-sur-Seine
  - Research Site, Jarny
  - Research Site, Jarville-la-Malgrange
  - Research Site, Jassans-Riottier
  - Research Site, Jonquières-Saint-Vincent
  - Research Site, Joué-lès-Tours
  - Research Site, Jouy-le-Châtel
  - Research Site, Juan-les-Pins
  - Research Site, Jœuf
  - Research Site, Kédange-sur-Canner
  - Research Site, L'Isle-d'Abeau
  - Research Site, La Baule-Escoublac
  - Research Site, La Chapelle-d'Angillon
  - Research Site, La Chapelle-en-Serval
  - Research Site, La Chapelle-la-Reine
  - Research Site, La Courneuve
  - Research Site, La Côte-Saint-André
  - Research Site, La Destrousse
  - Research Site, La Ferté-Milon
  - Research Site, La Ferté-Saint-Aubin
  - Research Site, La Ferté-sous-Jouarre
  - Research Site, La Fère
  - Research Site, La Fouillade
  - Research Site, La Frette-sur-Seine
  - Research Site, La Garde
  - Research Site, La Garnache
  - Research Site, La Haye-du-Puits
  - Research Site, La Haye-Pesnel
  - Research Site, La Mulatière
  - Research Site, La Neuville-Roy
  - Research Site, La Primaube
  - Research Site, La Queue-en-Brie
  - Research Site, La Réole
  - Research Site, La Rivière-Saint-Sauveur
  - Research Site, La Rochelle
  - Research Site, La Seyne-sur-Mer
  - Research Site, La Source
  - Research Site, La Trimouille
  - Research Site, La Tronche
  - Research Site, La Valette-du-Var
  - Research Site, Labenne
  - Research Site, Labruguière
  - Research Site, Lacapelle-Biron
  - Research Site, Lachapelle-aux-Pots
  - Research Site, Lamagistère
  - Research Site, Lambersart
  - Research Site, Lamorlaye
  - Research Site, Lamotte-Beuvron
  - Research Site, Landes
  - Research Site, Landivisiau
  - Research Site, Landouge
  - Research Site, Lannion
  - Research Site, Lanvallay
  - Research Site, Lanvéoc
  - Research Site, Laon
  - Research Site, Lapugnoy
  - Research Site, Largentière
  - Research Site, Larmor-Plage
  - Research Site, Laudun-lArdoise
  - Research Site, Lavardac
  - Research Site, Laveline-devant-Bruyères
  - Research Site, Lavoncourt
  - Research Site, Le Blanc-Mesnil
  - Research Site, Le Bourg-d'Oisans
  - Research Site, Le Bourget
  - Research Site, Le Bourget-du-Lac
  - Research Site, Le Bouscat
  - Research Site, Le Breuil-en-Auge
  - Research Site, Le Brusc
  - Research Site, Le Cannet
  - Research Site, Le Creusot
  - Research Site, Le Golfe Juan
  - Research Site, Le Grand-Lemps
  - Research Site, Le Grau-du-Roi
  - Research Site, Le Havre
  - Research Site, Le Kremlin-Bicêtre
  - Research Site, Le Lavandou
  - Research Site, Le Lude
  - Research Site, Le Mans
  - Research Site, Le Neubourg
  - Research Site, Le Pertre
  - Research Site, Le Petit Clamart
  - Research Site, Le Pin
  - Research Site, Le Plessis-Bouchard
  - Research Site, Le Pontet
  - Research Site, Le Puy-en-Velay
  - Research Site, Le Relecq-Kerhuon
  - Research Site, Le Rove
  - Research Site, Le Sequestre
  - Research Site, Le Soler
  - Research Site, Le Teil
  - Research Site, Le Temple-de-Bretagne
  - Research Site, Le Thor
  - Research Site, Le Tréport
  - Research Site, Le Val-dAjol
  - Research Site, Lecci
  - Research Site, Lembach
  - Research Site, Lens
  - Research Site, Les Abrets
  - Research Site, Les Issambres
  - Research Site, Les Mées
  - Research Site, Les Milles
  - Research Site, Les Mureaux
  - Research Site, Les Pavillons-sous-Bois
  - Research Site, Les Pujols
  - Research Site, Les Sables-d'Olonne
  - Research Site, Lescheraines
  - Research Site, Lesparre-Médoc
  - Research Site, Levallois-Perret
  - Research Site, Leyme
  - Research Site, Lezoux
  - Research Site, Lézardrieux
  - Research Site, Lézignan-Corbières
  - Research Site, Liffré
  - Research Site, Ligny-en-Barrois
  - Research Site, Ligny-en-Cambrésis
  - Research Site, Lille
  - Research Site, Lillebonne
  - Research Site, Limoges
  - Research Site, Lingolsheim
  - Research Site, Livry-Gargan
  - Research Site, Lognes
  - Research Site, Lombez
  - Research Site, Lomme
  - Research Site, Longueau
  - Research Site, Longué-Jumelles
  - Research Site, Lons-le-Saunier
  - Research Site, Lormont
  - Research Site, Louverné
  - Research Site, Louvigné-de-Bais
  - Research Site, Louvigné-du-Désert
  - Research Site, Luçon
  - Research Site, Lunel
  - Research Site, Lunéville
  - Research Site, Luxeuil-les-Bains
  - Research Site, Lyon
  - Research Site, Lys-lez-Lannoy
  - Research Site, Magalas
  - Research Site, Maintenon
  - Research Site, Mainvilliers
  - Research Site, Maisons-Alfort
  - Research Site, Malaucène
  - Research Site, Malemort-sur-Corrèze
  - Research Site, Mandeure
  - Research Site, Manduel
  - Research Site, Manosque
  - Research Site, Mantes-la-Ville
  - Research Site, Marcilloles
  - Research Site, Marcq-en-Barœul
  - Research Site, Mareuil-sur-Lay-Dissais
  - Research Site, Margency
  - Research Site, Marguerittes
  - Research Site, Marignane
  - Research Site, Marle
  - Research Site, Marlenheim
  - Research Site, Marles-les-Mines
  - Research Site, Marmande
  - Research Site, Maromme
  - Research Site, Marquette-lez-Lille
  - Research Site, Marquillies
  - Research Site, Marquion
  - Research Site, Marsannay-la-Côte
  - Research Site, Marseille
  - Research Site, Marspich
  - Research Site, Martigues
  - Research Site, Marvejols
  - Research Site, Mas-Grenier
  - Research Site, Masseret
  - Research Site, Massy
  - Research Site, Matha
  - Research Site, Maubeuge
  - Research Site, Mauguio
  - Research Site, Maule
  - Research Site, Mauléon-Licharre
  - Research Site, Maureillas-las-Illas
  - Research Site, Mauvezin
  - Research Site, Maxéville
  - Research Site, Mayenne
  - Research Site, Mennevret
  - Research Site, Menton
  - Research Site, Metz
  - Research Site, Meudon
  - Research Site, Meulan-en-Yvelines
  - Research Site, Meursault
  - Research Site, Meusnes
  - Research Site, Meyzieu
  - Research Site, Mezel
  - Research Site, Méjannes-lès-Alès
  - Research Site, Mériel
  - Research Site, Mérindol
  - Research Site, Méru
  - Research Site, Mézidon-Canon
  - Research Site, Mézières-en-Brenne
  - Research Site, Mézy-sur-Seine
  - Research Site, Migennes
  - Research Site, Milhaud
  - Research Site, Millau
  - Research Site, Mimizan
  - Research Site, Miramas
  - Research Site, Miramont-de-Guyenne
  - Research Site, Mirecourt
  - Research Site, Mitry-Mory
  - Research Site, Mittelhausen
  - Research Site, Mittersheim
  - Research Site, Moissy-Cramayel
  - Research Site, Molsheim
  - Research Site, Moncé-en-Belin
  - Research Site, Monéteau
  - Research Site, Monswiller
  - Research Site, Montauban
  - Research Site, Montceau-les-Mines
  - Research Site, Montchanin
  - Research Site, Montcy-Notre-Dame
  - Research Site, Montdidier
  - Research Site, Montereau-Fault-Yonne
  - Research Site, Montesson
  - Research Site, Monteux
  - Research Site, Montélimar
  - Research Site, Montévrain
  - Research Site, Montigny-le-Roi
  - Research Site, Montigny-lès-Metz
  - Research Site, Montluçon
  - Research Site, Montmagny
  - Research Site, Montmorillon
  - Research Site, Montoire-sur-le-Loir
  - Research Site, Montpellier
  - Research Site, Montreuil
  - Research Site, Montreuil-Bellay
  - Research Site, Montréal
  - Research Site, Montrouge
  - Research Site, Morcenx
  - Research Site, Moreuil
  - Research Site, Morhange
  - Research Site, Morlaix
  - Research Site, Mortagne-du-Nord
  - Research Site, Mortain
  - Research Site, Mougins
  - Research Site, Mouriès
  - Research Site, Moussey
  - Research Site, Mouy
  - Research Site, Moyeuvre-Grande
  - Research Site, Mundolsheim
  - Research Site, Muret
  - Research Site, Naintré
  - Research Site, Nançay
  - Research Site, Nanterre
  - Research Site, Nantes
  - Research Site, Nantua
  - Research Site, Narbonne
  - Research Site, Naucelle
  - Research Site, Neauphle-le-Château
  - Research Site, Nemours
  - Research Site, Neufchef
  - Research Site, Neuilly-le-Réal
  - Research Site, Neuilly-lès-Dijon
  - Research Site, Neuville-lès-Dieppe
  - Research Site, Nexon
  - Research Site, Nice
  - Research Site, Nielles-lès-Bléquin
  - Research Site, Niort
  - Research Site, Nîmes
  - Research Site, Nogent-le-Phaye
  - Research Site, Nogent-le-Roi
  - Research Site, Nogent-le-Rotrou
  - Research Site, Noirmoutier-en-l'Île
  - Research Site, Noisy-le-Grand
  - Research Site, Noisy-le-Sec
  - Research Site, Nomain
  - Research Site, Notre-Dame-de-Gravenchon
  - Research Site, Nouâtre
  - Research Site, Noyers-sur-Cher
  - Research Site, Noyon
  - Research Site, Nœux-les-Mines
  - Research Site, Oberhausbergen
  - Research Site, Obernai
  - Research Site, Oinville-sur-Montcient
  - Research Site, Oisemont
  - Research Site, Oisseau
  - Research Site, Olby
  - Research Site, Olivet
  - Research Site, Orange
  - Research Site, Orchies
  - Research Site, Orléans
  - Research Site, Orly
  - Research Site, Ormes
  - Research Site, Orry-la-Ville
  - Research Site, Orthez
  - Research Site, Orvault
  - Research Site, Oudon
  - Research Site, Oullins
  - Research Site, Oyonnax
  - Research Site, Ozoir-la-Ferrière
  - Research Site, Pagny-sur-Moselle
  - Research Site, Paimpol
  - Research Site, Pantin
  - Research Site, Parcey
  - Research Site, Parempuyre
  - Research Site, Paris
  - Research Site, Passavant-la-Rochère
  - Research Site, Passy
  - Research Site, Pau
  - Research Site, Perpignan
  - Research Site, Perreux
  - Research Site, Petite-Synthe
  - Research Site, Périgueux
  - Research Site, Pibrac
  - Research Site, Pierrepont-sur-Avre
  - Research Site, Pins-Justaret
  - Research Site, Pipriac
  - Research Site, Pisany
  - Research Site, Plaimpied-Givaudins
  - Research Site, Plaisance
  - Research Site, Plaisance-du-Touch
  - Research Site, Plan-de-Cuques
  - Research Site, Plancher-les-Mines
  - Research Site, Pleaux
  - Research Site, Plessala
  - Research Site, Plestin-les-Grèves
  - Research Site, Pleumeur-Gautier
  - Research Site, Pléhédel
  - Research Site, Ploemeur
  - Research Site, Plombières-lès-Dijon
  - Research Site, Plouescat
  - Research Site, Plouguernével
  - Research Site, Plourhan
  - Research Site, Plouzané
  - Research Site, Pluméliau
  - Research Site, Poitiers
  - Research Site, Poncin
  - Research Site, Pont-à-Mousson
  - Research Site, Pont-Évêque
  - Research Site, Pont-l'Abbé-d'Arnoult
  - Research Site, Pontcharra
  - Research Site, Ponte Leccia
  - Research Site, Pornic
  - Research Site, Port-Saint-Louis-du-Rhône
  - Research Site, Port-sur-Saône
  - Research Site, Portet-sur-Garonne
  - Research Site, Potigny
  - Research Site, Pouilley-les-Vignes
  - Research Site, Pouilly-en-Auxois
  - Research Site, Poulx
  - Research Site, Pré-en-Pail
  - Research Site, Prigonrieux
  - Research Site, Privas
  - Research Site, Prunelli Di Fium Orbo
  - Research Site, Puget-Ville
  - Research Site, Puichéric
  - Research Site, Pulnoy
  - Research Site, Puteaux
  - Research Site, Puttelange-aux-Lacs
  - Research Site, Puy-lÉvêque
  - Research Site, Questembert
  - Research Site, Quevauvillers
  - Research Site, Quincy-sous-Sénart
  - Research Site, Quincy-Voisins
  - Research Site, Rambervillers
  - Research Site, Ramonville-Saint-Agne
  - Research Site, Râches
  - Research Site, Rebais
  - Research Site, Redon
  - Research Site, Rennes
  - Research Site, Ribemont
  - Research Site, Richardménil
  - Research Site, Rieumes
  - Research Site, Rieupeyroux
  - Research Site, Rieux
  - Research Site, Rillieux-la-Pape
  - Research Site, Riom
  - Research Site, Riquewihr
  - Research Site, Rixheim
  - Research Site, Roanne
  - Research Site, Roche-la-Molière
  - Research Site, Rochefort
  - Research Site, Rodez
  - Research Site, Rognac
  - Research Site, Rohrbach-lès-Bitche
  - Research Site, Roissy-en-Brie
  - Research Site, Roissy-en-France
  - Research Site, Rombas
  - Research Site, Roncey
  - Research Site, Roncq
  - Research Site, Roquebrune-Cap-Martin
  - Research Site, Roubaix
  - Research Site, Rouen
  - Research Site, Rouhling
  - Research Site, Rouillé
  - Research Site, Roulans
  - Research Site, Royan
  - Research Site, Roye
  - Research Site, Rue
  - Research Site, Rugles
  - Research Site, Sabres
  - Research Site, Sains-du-Nord
  - Research Site, Saint Marc Sur Mer
  - Research Site, Saint Maximin La Ste Baume
  - Research Site, Saint-Amand-sur-Fion
  - Research Site, Saint-Amé
  - Research Site, Saint-Amour
  - Research Site, Saint-André-de-Sangonis
  - Research Site, Saint-André-des-Eaux
  - Research Site, Saint-André-lez-Lille
  - Research Site, Saint-Arnoult-en-Yvelines
  - Research Site, Saint-Aubert
  - Research Site, Saint-Avertin
  - Research Site, Saint-Barthélemy-de-Vals
  - Research Site, Saint-Benoît
  - Research Site, Saint-Branchs
  - Research Site, Saint-Brice-sous-Forêt
  - Research Site, Saint-Ciers-sur-Gironde
  - Research Site, Saint-Cyr-sur-Loire
  - Research Site, Saint-Denis
  - Research Site, Saint-Denis-dAnjou
  - Research Site, Saint-Erme-Outre-et-Ramecourt
  - Research Site, Saint-Estève
  - Research Site, Saint-Etienne
  - Research Site, Saint-Égrève
  - Research Site, Saint-Félix-de-Lodez
  - Research Site, Saint-Flour
  - Research Site, Saint-Gaudens
  - Research Site, Saint-Germain-du-Plain
  - Research Site, Saint-Germain-du-Puch
  - Research Site, Saint-Germain-en-Laye
  - Research Site, Saint-Germain-Laval
  - Research Site, Saint-Germainmont
  - Research Site, Saint-Gratien
  - Research Site, Saint-Herblain
  - Research Site, Saint-Hilaire-lez-Cambrai
  - Research Site, Saint-Jacques-sur-Darnétal
  - Research Site, Saint-Jean-de-la-Ruelle
  - Research Site, Saint-Jean-de-Monts
  - Research Site, Saint-Jean-des-Baisants
  - Research Site, Saint-Jorioz
  - Research Site, Saint-Julien-sur-Cher
  - Research Site, Saint-Just-Saint-Rambert
  - Research Site, Saint-Laurent-d'Aigouze
  - Research Site, Saint-Laurent-du-Var
  - Research Site, Saint-Léger-en-Yvelines
  - Research Site, Saint-Léger-sous-Cholet
  - Research Site, Saint-Loubès
  - Research Site, Saint-Marcel-Bel-Accueil
  - Research Site, Saint-Martin-Boulogne
  - Research Site, Saint-Martin-des-Champs
  - Research Site, Saint-Mathieu-de-Tréviers
  - Research Site, Saint-Maurice-sur-Moselle
  - Research Site, Saint-Médard-d'Eyrans
  - Research Site, Saint-Nicolas-de-Port
  - Research Site, Saint-Omer
  - Research Site, Saint-Paul-Trois-Châteaux
  - Research Site, Saint-Pierre-des-Corps
  - Research Site, Saint-Priest
  - Research Site, Saint-Priest-en-Jarez
  - Research Site, Saint-Quentin
  - Research Site, Saint-Quentin-la-Poterie
  - Research Site, Saint-Rambert-d'Albon
  - Research Site, Saint-Raphaël
  - Research Site, Saint-Rémy-de-Provence
  - Research Site, Saint-Saëns
  - Research Site, Saint-Saulve
  - Research Site, Saint-Sauveur-dAunis
  - Research Site, Saint-Sauveur-le-Vicomte
  - Research Site, Saint-Savinien
  - Research Site, Saint-Sébastien-sur-Loire
  - Research Site, Saint-Thibéry
  - Research Site, Saint-Thuriau
  - Research Site, Saint-Urbain
  - Research Site, Saint-Vallier
  - Research Site, Saint-Vrain
  - Research Site, Saintes
  - Research Site, Salles
  - Research Site, Sanary-sur-Mer
  - Research Site, Sargé-lès-le-Mans
  - Research Site, Sarlat-la-Canéda
  - Research Site, Sarrebourg
  - Research Site, Sarry
  - Research Site, Sartrouville
  - Research Site, Sault-lès-Rethel
  - Research Site, Saulxures-lès-Nancy
  - Research Site, Sauveterre-de-Béarn
  - Research Site, Saverne
  - Research Site, Savignac-les-Églises
  - Research Site, Savigny-le-Temple
  - Research Site, Savigny-sur-Orge
  - Research Site, Savonnières
  - Research Site, Scey-sur-Saône-et-Saint-Albin
  - Research Site, Schiltigheim
  - Research Site, Sedan
  - Research Site, Segonzac
  - Research Site, Seichamps
  - Research Site, Sens
  - Research Site, Sens-de-Bretagne
  - Research Site, Seraincourt
  - Research Site, Seveux
  - Research Site, Seyssinet-Pariset
  - Research Site, Seyssuel
  - Research Site, Sète
  - Research Site, Sélestat
  - Research Site, Séméac
  - Research Site, Sérignan
  - Research Site, Sillé-le-Guillaume
  - Research Site, Simiane-Collongue
  - Research Site, Sochaux
  - Research Site, Soissons
  - Research Site, Solliès-Pont
  - Research Site, Solre-le-Château
  - Research Site, Sonchamp
  - Research Site, Sorgues
  - Research Site, Soufflenheim
  - Research Site, Souillac
  - Research Site, Soyaux
  - Research Site, Ste Florine
  - Research Site, Ste Luce Sur Loire
  - Research Site, Ste Menehould
  - Research Site, Strasbourg
  - Research Site, Suresnes
  - Research Site, Tarbes
  - Research Site, Tartas
  - Research Site, Tassin-la-Demi-Lune
  - Research Site, Teloché
  - Research Site, Templeuve-en-Pévèle
  - Research Site, Tence
  - Research Site, Téteghem
  - Research Site, Thann
  - Research Site, Théoule-sur-Mer
  - Research Site, Thiberville
  - Research Site, Thilouze
  - Research Site, Thoirette
  - Research Site, Thorigné-sur-Dué
  - Research Site, Thouaré-sur-Loire
  - Research Site, Thouars
  - Research Site, Thuir
  - Research Site, Thun-Saint-Amand
  - Research Site, Til-Châtel
  - Research Site, Tilly-sur-Seulles
  - Research Site, Tonnay-Boutonne
  - Research Site, Tonneins
  - Research Site, Torcy
  - Research Site, Toul
  - Research Site, Toulon
  - Research Site, Touques
  - Research Site, Tourcoing
  - Research Site, Tournefeuille
  - Research Site, Tours
  - Research Site, Tourves
  - Research Site, Tracy-le-Mont
  - Research Site, Traînel
  - Research Site, Trangé
  - Research Site, Trévières
  - Research Site, Trie-sur-Baïse
  - Research Site, Uckange
  - Research Site, Ury
  - Research Site, Ussac
  - Research Site, Ussel
  - Research Site, Vailly-sur-Aisne
  - Research Site, Valbonne
  - Research Site, Valence
  - Research Site, Valenciennes
  - Research Site, Valff
  - Research Site, Vals-les-Bains
  - Research Site, Vandœuvre-lès-Nancy
  - Research Site, Varces-Allières-et-Risset
  - Research Site, Varennes-Jarcy
  - Research Site, Vasles
  - Research Site, Vaulnaveys-le-Haut
  - Research Site, Vaulx-en-Velin
  - Research Site, Vaux-le-Pénil
  - Research Site, Veigné
  - Research Site, Venarey-les-Laumes
  - Research Site, Vendôme
  - Research Site, Verneuil-sur-Avre
  - Research Site, Verneuil-sur-Seine
  - Research Site, Vernouillet
  - Research Site, Verquières
  - Research Site, Versailles
  - Research Site, Vertaizon
  - Research Site, Verton
  - Research Site, Vervins
  - Research Site, Vélizy-Villacoublay
  - Research Site, Vénissieux
  - Research Site, Vétheuil
  - Research Site, Vic-la-Gardiole
  - Research Site, Vichy
  - Research Site, Vienne
  - Research Site, Vierzon
  - Research Site, Vieugy
  - Research Site, Vigoulet
  - Research Site, Villars-les-Dombes
  - Research Site, Villeblevin
  - Research Site, Villedieu-sur-Indre
  - Research Site, Villefranche-de-Lonchat
  - Research Site, Villefranche-sur-Saône
  - Research Site, Villejuif
  - Research Site, Villemoisson-sur-Orge
  - Research Site, Villeneuve-d'Ascq
  - Research Site, Villeneuve-la-Garenne
  - Research Site, Villeneuve-le-Roi
  - Research Site, Villeneuve-lès-Avignon
  - Research Site, Villepreux
  - Research Site, Villers-Bretonneux
  - Research Site, Villerupt
  - Research Site, Villeurbanne
  - Research Site, Villevocance
  - Research Site, Vimy
  - Research Site, Vinay
  - Research Site, Vincennes
  - Research Site, Vitrolles
  - Research Site, Vitry-le-François
  - Research Site, Vitry-sur-Orne
  - Research Site, Vitry-sur-Seine
  - Research Site, Vittel
  - Research Site, Vivy
  - Research Site, Vizille
  - Research Site, Voiron
  - Research Site, Voisins-le-Bretonneux
  - Research Site, Vonnas
  - Research Site, Vouillé
  - Research Site, Voujeaucourt
  - Research Site, Walincourt-Selvigny
  - Research Site, Wambrechies
  - Research Site, Warmeriville
  - Research Site, Wasquehal
  - Research Site, Wasselonne
  - Research Site, Wattrelos
  - Research Site, Waziers
  - Research Site, Witry-lès-Reims
  - Research Site, Wittelsheim
  - Research Site, Woippy
  - Research Site, Yvetot
  - Research Site, Yvré-le-Pôlin